CLINICAL TRIAL: NCT06067399
Title: Relationship Between Red Cell Distribution Width (RDW) and HbA1C in Patients With Type 2 Diabetes Mellitus After Glycemic Control
Status: Recruiting | Type: Observational
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer of Internal Medicine and Clinical Hematology, New Valley University
Other Study IDs: T2DMRDW
Record Dates: First submitted 2023-09-21; First posted 2023-10-04 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Diabetics
  Interventions: Diagnostic Test: Glycated hemoglobin (HbA1C); Diagnostic Test: RDW; Diagnostic Test: Lipid profile
- 2: Healthy control
  Interventions: Diagnostic Test: Glycated hemoglobin (HbA1C); Diagnostic Test: RDW; Diagnostic Test: Lipid profile

INTERVENTIONS:
Diagnostic Test: Glycated hemoglobin (HbA1C) — Blood test will be done at time of recruitment (for 2 groups) , after 3 months and after 6 months (for group 1 )
Diagnostic Test: RDW — Blood test will be done at time of recruitment (for 2 groups) , after 3 months and after 6 months (for group 1 )
Diagnostic Test: Lipid profile — Blood test will be done at time of recruitment (for 2 groups) , after 3 months and after 6 months (for group 1 )

SUMMARY:
Diabetes mellitus (DM) is an epidemic disease, with approximately 463 million persons diagnosed with it. Of those, 90% are patients with type 2 DM (T2DM). Some estimates indicate that 700 million cases of DM will be reported in 2045. T2DM develops due to insulin resistance, leading to reduced insulin secretion. DM has a number of associated complications, such as nephropathy, neuropathy, and cardiovascular disease.

DETAILED DESCRIPTION:
The health status of normal individuals and patients with various diseases is commonly monitored using the complete blood count (CBC). In patients with T2DM, the CBC can be used as a follow-up test, which will help in reducing complications associated with the disease. Some CBC parameters have also been used as prognostic markers for T2DM. One of these markers is the red cell distribution width (RDW), which measures the variability in the sizes of red blood cells (RBCs) and is considered an indicator of their heterogeneity. The evidence associating RDW with a higher risk of mortality has been expanding since the initial report of its prognostic utility in heart failure patients. Multiple studies have shown that elevated RDW values are associated with many human diseases, such as cancer, cardiovascular disease, and diabetes, and are also associated with disease activity or complications of diseases. The RDW can be used diagnostically in patients with T2DM and other illnesses, as patients with T2DM frequently show alterations in various hematological properties, including changes in the structure, metabolism, and function of blood cells. These alterations can be caused by different factors, such as excessive levels of reactive oxygen species (ROS), leading eventually to oxidative stress and the dysfunction of RBCs.

The relationship between RDW and T2DM has been studied for several years, and there are no consistent results.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have Uncontrolled type 2 diabetes mellitus (HbA1C more than 7%)

Exclusion Criteria:

1. Patients diagnosed to have type 1 diabetes.
2. Patients are diagnosed to have secondary diabetes.
3. Clinical states associated with increased RDW:

   * Anemia (Female Hb less than 12, Male Hb less than 13) either due to hemolysis, or in response to ineffective red cell production, which can be caused by deficiencies in iron, vitamin B12 or folate.
   * After blood transfusions
   * Pregnancy, thrombotic thrombocytopenic purpura and inflammatory bowel disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed to have type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the correlation between RDW and HbA1C levels in patients with T2DM before and after glycemic control. | "At time of inclusion in the study", "3 months", "6 months"

SECONDARY OUTCOMES:
To determine if changes in RDW levels correlate with the presence of other comorbidities and complications. | once

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University- Faculty of Medicine, Al Khārjah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valtierra-Alvarado MA, Castaneda Delgado JE, Ramirez-Talavera SI, Lugo-Villarino G, Duenas-Arteaga F, Lugo-Sanchez A, Adame-Villalpando MS, Rivas-Santiago B, Enciso-Moreno J, Serrano CJ. Type 2 diabetes mellitus metabolic control correlates with the phenotype of human monocytes and monocyte-derived macrophages. J Diabetes Complications. 2020 Nov;34(11):107708. doi: 10.1016/j.jdiacomp.2020.107708. Epub 2020 Aug 13. PMID 32843282
- [Background] Ooi TC, Mat Ludin AF, Loke SC, Fiatarone Singh MA, Wong TW, Vytialingam N, Anthony Abdullah MMJ, Ng OC, Bahar N, Zainudin N, Lew LC. A 16-Week Home-Based Progressive Resistance Tube Training Among Older Adults With Type-2 Diabetes Mellitus: Effect on Glycemic Control. Gerontol Geriatr Med. 2021 Aug 12;7:23337214211038789. doi: 10.1177/23337214211038789. eCollection 2021 Jan-Dec. PMID 34409130
- [Background] Nah EH, Cho S, Park H, Kim S, Cho HI. Associations of complete blood count parameters with pancreatic beta-cell function and insulin resistance in prediabetes and type 2 diabetes mellitus. J Clin Lab Anal. 2022 Jun;36(6):e24454. doi: 10.1002/jcla.24454. Epub 2022 May 13. PMID 35561266
- [Background] Bhutto AR, Abbasi A, Abro AH. Correlation of Hemoglobin A1c with Red Cell Width Distribution and Other Parameters of Red Blood Cells in Type II Diabetes Mellitus. Cureus. 2019 Aug 30;11(8):e5533. doi: 10.7759/cureus.5533. PMID 31687307
- [Background] Arkew M, Yemane T, Mengistu Y, Gemechu K, Tesfaye G. Hematological parameters of type 2 diabetic adult patients at Debre Berhan Referral Hospital, Northeast Ethiopia: A comparative cross-sectional study. PLoS One. 2021 Jun 14;16(6):e0253286. doi: 10.1371/journal.pone.0253286. eCollection 2021. PMID 34125859